CLINICAL TRIAL: NCT05004194
Title: Vestibular Caloric Stimulation and the Modulation of Pain in Fibromyalgia: An Open Label Pilot Study
Brief Title: Vestibular Caloric Stimulation and the Modulation of Pain in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ioannis Tassiulas, Associate Professor of Medicine, Rheumatology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-2730
Record Dates: First submitted 2021-08-09; First posted 2021-08-13 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: An open label non-randomized pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cold water caloric stimulation (Experimental): 50 cc of ice-cold water irrigation into the right ear at 1-2 cc/second, once per participant.
  Interventions: Procedure: Vestibular Caloric Stimulation

INTERVENTIONS:
Procedure: Vestibular Caloric Stimulation — Irrigation of the right external ear canal
  Other Names: VCS; Cold water caloric stimulation

SUMMARY:
The management of chronic pains is challenging and fraught with limitations. Fibromyalgia is a common pain disorder characterized by chronic widespread pains, associated with fatigue and impaired quality of life. Fibromyalgia affects millions of people and is among the most common reasons for consulting with a rheumatologist. The food and drug administration (FDA) approved three medications to treat fibromyalgia, though there are many patients for whom these medications are ineffective, poorly tolerated or cost-prohibitive. Accordingly, there exists a need for novel therapeutics.

The researchers would like to test the therapeutic efficacy of a non-pharmacologic non-interventional bedside technique called vestibular caloric stimulation (VCS). VCS, irrigating the external ear canal with water, is a simple, non-invasive, cost-free procedure with preliminary data suggesting potential for improving pain. VCS is a form of neuromodulation and there are anatomically defined pathways elucidated to help explain how this works. There currently exists limited data on the topic, only case reports and case series. Given a clear need for additional therapeutics in many patients with fibromyalgia, the researchers have elected to conduct this trial.

DETAILED DESCRIPTION:
This is an open label pilot study testing the potential therapeutic efficacy of vestibulocortical stimulation via cold water calorics in fibromyalgia. The trial will entail 6 weeks of total involvement for each participant including 3 weeks of active participation, with 4 weeks follow up: the irrigation happens at the beginning of week 2, so 4 weeks later is week 6.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old with ability to comprehend and consent to protocol.
* Diagnosis of fibromyalgia by American College of Rheumatology (ACR) criteria (questionnaire).
* At least a 4/10 baseline on the visual analogue pain scale (VAS).
* Stable fibromyalgia medications for at least 4 weeks.
* Owns or has access to a smart phone or computer to complete outcome measures.

Exclusion Criteria:

* Use of opioids
* Otitis externa or media within the past six months.
* Current ear pain with or without other symptoms of otitis externa.
* History of tympanic membrane rupture or surgery.
* Current pregnancy.
* Inability to lay supine for 30 minutes.
* Limited decision making capacity.
* Engaged in litigation, currently or prior, related to FMS.
* Inability to commute to clinic once.
* Primary language not English.
* Clinically significant or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise participation in the study
* Treatment with the medication meclizine for vertigo
* History of seizures
* Diagnosis of bipolar disorder (treated or untreated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Rating Scale (NRS) | baseline and 1 week after VCS
  Change in average diary pain scores assessed by daily report on a 11 point numeric rating scale at 1 week after VCS as compared to baseline. Full scale range from 0-10, higher score indicates more pain.

SECONDARY OUTCOMES:
Acute change in NRS | baseline and 5, 15 and 30 minutes after VCS
  Acute effect of VCS assessed by acute change in pain scores post VCS 5, 15 and 30 minutes post irrigation compared to baseline. Full scale range from 0-10, higher score indicates more pain.
Percentage of participants with NRS pain scores >= to 30% and 50% | 30 minutes, 24 hours, 1 week, 2 weeks after VCS
  Percentage of patients with change in pain assessed by NRS pain scores > or equal to 30% and 50%.
Patient Global Impression of Change (PGIC) | at 1 weeks, 2 weeks and 4 weeks after VCS
  Full score from 0-7, with higher score indicating more improvement.
Change in Multidimensional Assessment of Fatigue (MAF) | baseline and at 1, 2 and 4 weeks after VCS
  MAF is a 16 item instrument, full scale from 0-50, with higher score indicating more fatigue.
Michigan Neuropathy Screening Instrument (MNSI) | baseline and at 1, 2 and 4 weeks after VCS
  15 "yes or no" questions - full score from 0-13, with higher score indicating more neuropathic symptoms.
Change in Brief Pain Inventory Short Form 36 (BPI SF36) | baseline and at 24 hours, 1 week, 2 weeks, 4 weeks after VCS
  A 9-item instrument with total score from 0 to 10, with higher score indicating worse outcomes. Will exclude question 2 which is a diagram and question 7 which asks about medications.
Change in Fibromyalgia Impact Questionnaire (FIQ) | baseline and at 1, 2 and 4 weeks after VCS
  Full scale from 0-100, with higher score indicating a greater impact of fibromyalgia syndrome.
Change in Numeric Rating Scale (NRS) for pain in different regions of the body | baseline and at 24 hours, 1 week, 2 week, 4 week after VCS
  Pain measured on a numeric rating scale in different regions of the body: the left upper extremity, right upper extremity, left lower extremity, right lower extremity, front of torso, back of torso, head/neck. Full scale range from 0-10, higher score indicates more pain.
VCS Tolerability Survey | 24 hours post VCS
  A seventeen question tolerability instrument developed specifically for caloric stimulation to assess tolerability by measuring the frequency and intensity of headaches, nausea, and vertigo. the tolerability scale does not have a total score just individual questions re headache nausea vertigo discomfort and grades intensities rated on a 0-10 scale, higher numbers reflecting higher severity of symptoms.
Number of participants willing to trial VCS again | 24 hours post VCS
  Number of participants expressing willingness to trial VCS again
Change in Subjective Overall Well Being Scale | at baseline and at 30 minutes after VCS, 24 hours, 1 week, 2 week and 4 weeks after VCS relative
  Subjective Overall Well Being Scale is a 11 point scale with full scale from 0-10, with higher score reflecting the best possible overall subjective disposition

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Tassiulas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No